CLINICAL TRIAL: NCT07104032
Title: A Phase 3, Multi-regional, Open-label, Randomized Study of Tirabrutinib vs Rituximab and Temozolomide in Participants With Relapsed/Refractory Primary Central Nervous System Lymphoma
Brief Title: Study of Tirabrutinib vs Rituximab/Temozolomide for Relapsed/Refractory Primary Central Nervous System Lymphoma (PCNSL)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Collaborators: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4059-17
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Relapsed/Refractory Primary Central Nervous System Lymphoma
Keywords: Bruton's tyrosine kinase (BTK)
MeSH Terms: conditions — Recurrence | interventions — tirabrutinib; Rituximab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirabrutinib (Experimental): Tirabrutinib 480 milligram (mg) orally every day (QD), as monotherapy in 28-day cycles.
  Interventions: Drug: Tirabrutinib
- Rituximab-Temozolomide (R-TMZ) (Active Comparator): Rituximab 375 milligram per square meter (mg/m2) intravenously (IV) and temozolomide 150 mg/m2/day orally, as combination therapy for Cycle 1 through 6.
  Interventions: Drug: Rituximab; Drug: Temozolomide

INTERVENTIONS:
Drug: Tirabrutinib — Administered orally.
  Other Names: ONO-4059
  Arms: Tirabrutinib
Drug: Rituximab — Administered intravenously (IV).
  Arms: Rituximab-Temozolomide (R-TMZ)
Drug: Temozolomide — Administered orally.
  Arms: Rituximab-Temozolomide (R-TMZ)

SUMMARY:
The purpose of this clinical trial is to evaluate efficacy and safety of tirabrutinib alone compared with rituximab and temozolomide (R-TMZ) combination therapy in participants with Relapsed/Refractory Primary Central Nervous System Lymphoma (PCNSL).

ELIGIBILITY:
Inclusion Criteria

1. Pathology report confirming the diagnosis of B-cell PCNSL
2. Relapsed or refractory B-cell PCNSL with at least 1 prior high-dose methotrexate (HD-MTX) based therapy for PCNSL:

   * Relapsed disease: Participants who achieved a response (CR, CRu, PR) to the last treatment and subsequently experienced disease progression.
   * Refractory disease: Participants whose best response to the last treatment was stable disease or PD.
3. One or more bi-dimensionally measurable brain lesions with a minimum diameter greater than or equal to (≥)1 centimeter (cm) × ≥1 cm in gadolinium-enhanced magnetic resonance imaging (MRI)
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2
5. Adequate bone marrow, renal, and hepatic function per central lab values
6. Participants must agree to comply with all defined contraceptive requirements

Exclusion Criteria

1. Participants with isolated intraocular PCNSL or spinal PCNSL with no brain lesions
2. Participants with non-B-cell PCNSL
3. Participants with systemic presence of lymphoma
4. Refractory to temozolomide with or without rituximab-containing regimens in the last PCNSL treatment
5. Concomitant systemic corticosteroid exposure within 14 days before starting study drug per Investigator assessment with the exception of the following:

   * Equivalent of up to 10 milligram per day (mg/day) of prednisone for a disease other than PCNSL
   * Equivalent of up to 50 mg/day of prednisone (equal to 8 mg/day dexamethasone) for participants with lesions of the brain and/or spinal cord
6. Active malignancy, other than PCNSL requiring systemic therapy
7. Poorly controlled comorbidity, or history of medical conditions contraindicated per Investigator assessment
8. Participants who are unable to swallow oral medication
9. Prior Bruton's tyrosine kinase inhibitor treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Estimated up to 24 months
  PFS based on blinded Independent Review Committee (BIRC) assessment according to International Primary Central Nervous System Lymphoma Collaborative Group (IPCG) criteria, defined as time from randomization to progressive disease (PD) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Estimated up to 48 months]
  ORR based on BIRC per IPCG criteria, defined as the percentage of participants with a best overall response of complete response (CR), unconfirmed complete response (CRu), or partial response (PR).
Overall Survival (OS) | Estimated up to 48 months
  OS defined as time from randomization until death due to any cause.
Complete Response Rate (CRR) | Estimated up to 48 months
  CRR based on BIRC per IPCG criteria, defined as the percentage of participants with a best overall response of CR or CRu.
Best Overall Response (BOR) | Estimated up to 48 months]
  BOR based on BIRC per IPCG criteria, defined as the best response from randomization to the date of PD or the date of initiation of subsequent anticancer therapy for PCNSL, whichever occurs first.
Time to Response (TTR) | Estimated up to 48 months
  TTR based on BIRC per IPCG criteria, defined as time between randomization and the date of first response of CR, CRu, or PR.
Time to Complete Response (TTCR) | Estimated up to 48 months
  TTCR based on BIRC per IPCG criteria, defined as the time between randomization and the date of first complete response (CR or CRu).
Duration of Response (DOR) | Estimated up to 48 months
  DOR based on BIRC per IPCG criteria, defined as the time between the date of first response (CR, CRu, or PR) and the date of the first PD or date of death due to any cause, whichever occurs first.
Disease Free Survival (DFS) | Estimated up to 48 months
  DFS based on BIRC per IPCG criteria, defined as the time between the date of first complete response (CR or CRu) and the date of the first PD, or date of death due to any cause, whichever occurs first.
Change from Baseline in Corticosteroid Dose | Baseline, estimated up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team, Study Director — Deciphera Pharmaceuticals, LLC
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No